CLINICAL TRIAL: NCT06190691
Title: An Open-label, Nonrandomized, Single-dose, Parallel-group, Safety, Tolerance, and Pharmacokinetic Study of LOXO-305 Administered to Fasted Hepatically Impaired Male and Female Subjects and Fasted Matched-control Healthy Subjects
Brief Title: Study of Pirtobrutinib (LOXO-305) in Participants With Impaired Liver Function and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20012; J2N-OX-JZNF (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pirtobrutinib (Normal Hepatic Function) (Experimental): Participants received a single dose of Pirtobrutinib 200 milligrams (mg) administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib (Mild Hepatic Impairment) (Experimental): Participants received a single dose of Pirtobrutinib 200 mg administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib (Moderate Hepatic Impairment) (Experimental): Participants received a single dose of Pirtobrutinib 200 mg administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib (Severe Hepatic Impairment) (Experimental): Participants received a single dose of Pirtobrutinib 200 mg administered orally on Day 1.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally
  Other Names: LOXO-305, LY3527727

SUMMARY:
The main purpose of this study is to measure how much of pirtobrutinib (LOXO-305) gets into the bloodstream and how long it takes the body to eliminate it in participants with impaired liver function and healthy participants. The side effects and tolerability of pirtobrutinib will also be evaluated. Participation could last about 46 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mild, moderate or severe hepatic impairment and healthy participants with normal hepatic function
* Males and females of non-childbearing potential.
* Within body mass index (BMI) range 18.5 to 40.0 kilograms per square meter (kg/m²).
* Participants will be in good health, based on medical history, physical examination findings, vital signs, 12 lead electrocardiogram (ECG), and clinical laboratory tests, as determined by the Investigator (or designee).
* Able to comply with all study procedures, including the 8-night stay at the Clinical Research Unit and follow-up phone call.

Exclusion Criteria:

* History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:

  1. pancreatitis
  2. peptic ulcer disease
  3. intestinal malabsorption
  4. gastric reduction surgery
  5. history or presence of clinically significant cardiovascular disease.
* Participants with out-of-range, at-rest vital signs.
* Abnormal laboratory values determined to be clinically significant by the Investigator (or designee).
* Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination.
* Participation in any other investigational study drug trial involving administration of any investigational drug in the past 30 days or 5 half-lives, whichever was longer, prior to the first dose administration (Day 1).
* Use or intention to use any prescription or over-the-counter medications within 14 days prior to the first dose administration (Day 1) and through end of trial.
* History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the participant at undue risk.
* Donation of blood from 56 days prior to Screening, plasma or platelets from 4 weeks prior to Screening.
* Receipt of blood products within 2 months prior to Check-in (Day -1).
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, biliary, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal (GI), neurological, or psychiatric disorder (as determined by the Investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renée Ward, MD, PhD, Study Director — Loxo Oncology
Locations (8):
- United States (8):
  - Orange County Research Institute, Anaheim, California
  - Orange County Research Center, Tustin, California
  - Riverside Clinical Research, Edgewater, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - Advanced Pharma Clinical Research, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirtobrutinib (Normal Hepatic Function); Pirtobrutinib (Moderate Hepatic Impairment); Pirtobrutinib (Severe Hepatic Impairment): Participants received a single dose of Pirtobrutinib 200 mg administered orally on Day 1.
- Pirtobrutinib (Mild Hepatic Impairment): Participants received a single dose of Pirtobrutinib 200 milligrams (mg) administered orally on Day 1.
Period: Overall Study
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Started | 14 | 8 | 8 | 6
Received Dose of Pirtobrutinib | 14 | 8 | 8 | 6
Completed | 12 | 8 | 8 | 6
Not Completed | 2 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment) | Total
Number analyzed (Participants) | 14 | 8 | 8 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (8.22) | 56.8 (4.560) | 56.3 (3.920) | 52.3 (9.350) | 55 (6.880)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 1 | 10
  Male | 10 | 5 | 6 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 4 | 5 | 19
  Not Hispanic or Latino | 9 | 3 | 4 | 1 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 0 | 0 | 5
  White | 11 | 6 | 8 | 6 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 8 | 8 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: All participants who received a dose of Pirtobrutinib, had at least 1 quantifiable plasma concentration of Pirtobrutinib and had at least 1 PK parameter computed. Subjects were excluded from the analysis if they experienced an AE of vomiting that occurred at or before 2 times the median Tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
nanogram per milliliter (ng/mL) | 4240 (32.4) | 4410 (22.7) | 4140 (20.8) | 3270 (22.8)

2. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: Tmax of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
hours | 2.50 [1 to 8] | 2.25 [1 to 6] | 2.25 [1 to 3] | 2.78 [2 to 4]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC0-t of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
hour*nanogram per milliliter (h*ng/mL) | 96800 (21.2) | 89900 (43) | 84600 (31.7) | 71500 (14.8)

4. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of Pirtobrutinib
Description: PK: AUC0-inf of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
hour*nanogram per milliliter (h*ng/mL) | 98000 (20.7) | 90900 (42.7) | 85700 (31.1) | 72200 (14.6)

5. Primary Outcome: PK: Percentage Extrapolation for AUC0-inf (%AUCextrap) of Pirtobrutinib
Description: PK: %AUCextrap of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
percentage of AUCextrap | 0.978 (67.3) | 1.13 (34.4) | 1.14 (54.7) | 0.921 (50.4)

6. Primary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t½) of Pirtobrutinib
Description: PK: t½ of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
hours | 21.2 (20.9) | 19.8 (27.7) | 18 (16.3) | 15.5 (26.6)

7. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Pirtobrutinib
Description: PK: CL/F of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
liter per hour (L/h) | 2.04 (20.7) | 2.20 (42.7) | 2.33 (31.1) | 2.77 (14.6)

8. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Pirtobrutinib
Description: PK: Vz/F of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
Liter (L) | 62.4 (29.5) | 62.9 (45.1) | 60.6 (30.1) | 61.8 (30.5)

9. Primary Outcome: PK: Mean Residence Time (MRT) of Pirtobrutinib
Description: MRT is the average time a drug molecule stays in the body, calculated from the AUC0-inf.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
hours | 28.8 (17.6) | 27.7 (26.3) | 25 (14) | 24 (26.2)

10. Primary Outcome: PK: Unbound Cmax (Cmax,u) of Pirtobrutinib
Description: Cmax,u was calculated by multiplying Cmax by Fu (i.e., Cmax*Fu). Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
nanogram per milliliter (ng/mL) | 107 (31.2) | 133 (16.3) | 118 (26.5) | 111 (27.5)

11. Primary Outcome: PK: Unbound AUC0-t (AUC0-t,u) of Pirtobrutinib
Description: AUC0-t,u was calculated by multiplying AUC0-t by Fu (i.e., AUC0-t*Fu). Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
hour*nanogram per milliliter (h*ng/mL) | 2440 (22.8) | 2710 (32.3) | 2410 (39.6) | 2410 (28.5)

12. Primary Outcome: PK: Unbound AUC0-inf (AUC0-inf,u) of Pirtobrutinib
Description: AUC0-inf,u was calculated by multiplying AUC0-inf by Fu (i.e., AUC0-inf*Fu). Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
hour*nanogram per milliliter (h*ng/mL) | 2470 (22.6) | 2740 (32.1) | 2440 (39.1) | 2440 (28.5)

13. Primary Outcome: PK: Unbound CL/F (CL/F,u) of Pirtobrutinib
Description: CL/F,u was calculated by multiplying CL/F by Fu (i.e., CL/F*Fu). Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
liter per hour (L/h) | 80.9 (22.6) | 73 (32.1) | 81.9 (39.1) | 82 (28.5)

14. Primary Outcome: PK: Unbound Vz/F (Vz/F,u) of Pirtobrutinib
Description: Vz/F,u was calculated by multiplying Vz/F by Fu (i.e., Vz/F*Fu). Fu represents the unbound fraction, which is the portion of the drug in the bloodstream that is unbound to plasma proteins. It is expressed as a decimal and will be calculated from protein binding concentration data as the unbound drug concentration divided by the total drug concentration in plasma. The concentrations of total and unbound drug were determined in a sample of predose plasma fortified with a known concentration of drug.
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 14 | 8 | 8 | 6
Liter (L) | 2470 (26) | 2090 (34) | 2130 (33.1) | 1830 (36.3)

15. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Normal Hepatic Function)
Description: PK: λZ of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Pirtobrutinib (Normal Hepatic Function)
Number analyzed (Participants) | 14
1/hour (1/h)
  Subject 1 | 0.0334
  Subject 2 | 0.0323
  Subject 3 | 0.0418
  Subject 4 | 0.0287
  Subject 5 | 0.0231
  Subject 6 | 0.0319
  Subject 7 | 0.0420
  Subject 8 | 0.0262
  Subject 9 | 0.0292
  Subject 10 | 0.0291
  Subject 11 | 0.0299
  Subject 12 | 0.0308
  Subject 13 | 0.0399
  Subject 14 | 0.0491

16. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Mild Hepatic Function)
Description: PK: λZ of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Pirtobrutinib (Mild Hepatic Impairment)
Number analyzed (Participants) | 8
1/hour (1/h)
  Subject 15 | 0.0270
  Subject 16 | 0.0448
  Subject 17 | 0.0453
  Subject 18 | 0.0336
  Subject 19 | 0.0234
  Subject 20 | 0.0273
  Subject 21 | 0.0432
  Subject 22 | 0.0440

17. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Moderate Hepatic Function)
Description: PK: λZ of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Pirtobrutinib (Moderate Hepatic Impairment)
Number analyzed (Participants) | 8
1/hour (1/h)
  Subject 23 | 0.0377
  Subject 24 | 0.0387
  Subject 25 | 0.0364
  Subject 26 | 0.0430
  Subject 27 | 0.0395
  Subject 28 | 0.0467
  Subject 29 | 0.0419
  Subject 30 | 0.0272

18. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib (Severe Hepatic Function)
Description: PK: λZ of pirtobrutinib
Time Frame: Day 1 (predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose)
Population: as for outcome 1
Measure: Number; unit: 1/hour (1/h)
Arm/Group | Pirtobrutinib (Severe Hepatic Impairment)
Number analyzed (Participants) | 6
1/hour (1/h)
  Subject 31 | 0.0401
  Subject 32 | 0.0526
  Subject 33 | 0.0279
  Subject 34 | 0.0522
  Subject 35 | 0.0465
  Subject 36 | 0.0567

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To Day 17)
Description: All participants who received a dose of Pirtobrutinib.
Arm/Group | Pirtobrutinib (Normal Hepatic Function) | Pirtobrutinib (Mild Hepatic Impairment) | Pirtobrutinib (Moderate Hepatic Impairment) | Pirtobrutinib (Severe Hepatic Impairment)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 3/14 | 2/8 | 0/8 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirtobrutinib (Normal Hepatic Function) (N=14) | Pirtobrutinib (Mild Hepatic Impairment) (N=8) | Pirtobrutinib (Moderate Hepatic Impairment) (N=8) | Pirtobrutinib (Severe Hepatic Impairment) (N=6)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT06190691/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT06190691/SAP_001.pdf